CLINICAL TRIAL: NCT03544801
Title: Renji Cerebral Small Vessel Disease Corhort Study
Acronym: RCCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: [2013012]
Record Dates: First submitted 2018-05-31; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Cerebrovascular Disorders; Cognition Disorders
MeSH Terms: conditions — Cerebrovascular Disorders; Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- sample group ,300: CSVD patients after symptomatic stroke
- control group,100: community population

SUMMARY:
We aim to make clear the impact with the mechanisms of variant pathological injuries on the outcomes of CSVD, to find independent imaging markers and establish prediction model of it.

DETAILED DESCRIPTION:
A cohort of post stroke cerebral small vessel disease (CSVD) patients with different cognitive status are consecutively recruited in this study. Detailed full domain cognitive assessment and multi-modal MRI (including brain morphology , DTI indices, microbleed counts, brain volumes as well as brain network characters, etc.) are performed. Cognitive states(including attention-executive function, memory, language, visuo-spatial and global cognition with the transition to dementia) and the overall prognosis (cardiovascular events, stroke recurrence, death due to cardiovascular event and all cause death) are longitudinally followed up. The correlations between baseline and followed MRI parameters with the outcomes are analyzed in order to make clear the impact with the mechanisms of variant pathological injuries on the outcomes of CSVD, to find independent imaging markers and establish prediction model of it.

ELIGIBILITY:
Inclusion Criteria:

* ①50-85 years; ② at least 6 years of education; ③ CSVD was defined as patients experienced a clinical lacunar stroke at least 1 months ago, and MRI showed responsible lacunar infarcts and white matter lesions; ④ Cooperate with cognitive tests; ⑤Not accept medications that affect cognition; ⑥. Score of modified Rankin scale ≦3; ⑦. Sign informed consent.

Exclusion Criteria:

* ① Etiology due to cardioembolic or large vessel disease (>50% stenosis in extra- or intra-cerebral arteries); ② Non vasular white matter lesions(WMLs)；③ Cortical and/or cortico-subcortical non-lacunar infarct; ④ Other cognitive diseases (such as Alzheimer's disease, Parkinson disease or thyroid disease, etc. ) ⑤Severe systemic diseases such as heart, liver and kidney diseases or major psychiatric disorders; ⑥Severe depressive state: Hamilton depression rating scale score >24; ⑦ MRI contraindications.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: longitudinal cohort of post stroke CSVD patients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-09-29 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
a predictive model | 2015,July---
  The occurrence, development and predictive imaging markers of cognitive impairment and overall outcomes in post stroke patients with cerebral small vessel diseases.

CONTACTS AND LOCATIONS:
Overall Officials: qun xu, professor, Study Chair — RenJi Hospital
Locations (1):
- Renji Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, China